CLINICAL TRIAL: NCT05483023
Title: 18-fluorofuranylnorprogesterone (FFNP) Positron Emission Tomography-Magnetic Resonance Imaging (PET/MRI) as a Potential Biomarker of Response to Progesterone Therapy in Complex Atypical Hyperplasia (CAH) and Grade 1 Endometrial Cancer (EC)
Brief Title: 18-fluorofuranylnorprogesterone (FFNP) PET/MRI as a Potential Biomarker of Response to Progesterone Therapy
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Drug cannot be produced and scanner down.
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Radiological Society of North America (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LCCC2221; 22-1677 (Other: UNC Chapel Hill IRB)
Record Dates: First submitted 2022-07-28; First posted 2022-08-01 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Complex Atypical Hyperplasia; Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 18F-fluorofuranylnorprogesterone PET / MRI (Experimental): All enrolled subjects will receive the tracer and then have a PET/MRI scan.
  Interventions: Drug: 18F-fluorofuranylnorprogesterone PET / MRI

INTERVENTIONS:
Drug: 18F-fluorofuranylnorprogesterone PET / MRI — Subjects will receive a PET/MRI with 18F-fluorofuranylnorprogesterone tracer

SUMMARY:
Purpose: The purpose of this study is to evaluate FFNP PET/MRI's utility for predicting response to Levonorgestrel-releasing Intrauterine Device (LR-IUD) hormonal therapy for Complex Atypical hyperplasia (CAH) and Endometrial Cancer (EC).

Participants: Eight women with histologically confirmed CAH or Grade 1 EC who have planned treatment with LR-IUD will be recruited..

Procedures (methods): The is a prospective, single arm, pilot study of 8 participants who will receive one FFNP PET/MRI scan. Medical records will be followed for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Female age 18 or older
* Histologically confirmed CAH or Grade 1 EC
* No prior surgical or hormonal treatment for CAH or Grade 1 EC
* Planned treatment with levonorgestrel-releasing intrauterine device (LR-IUD) for CAH or grade 1 EC

Exclusion Criteria:

* Inability to complete PET/MR scans due to severe claustrophobia
* Institutionalized subject (prisoner or nursing home subject)
* Implanted metallic devices, parts, vascular clips, or other foreign bodies.
* Known hypersensitivity to gadolinium or FFNP or to any component of gadolinium or FFNP refractory to standard medications (antihistamines, steroids)
* Impaired kidney function (serum creatinine level > 1.8 mg/dl or a glomerular filtration rate < 60 as approximated using serum creatinine levels) unless anuric and on dialysis.
* Any woman who is pregnant or has reason to believe she is pregnant (the possibility of pregnancy has to be excluded by negative urine (β-HCG) results, obtained within 24 hours before FFNP administration, or on the basis of patient history)
* Prior hormone treatment for breast cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Participant eligibility is based on the biological gender assigned at birth.
Enrollment: 0 (Actual)
Dates: Start 2024-02-15 (Actual); Primary Completion 2026-06-28 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of 18F-fluorofuranylnorprogesterone (FFNP) PET/MRI for predicting response to progestin therapy in CAH /EC patients | Upon completion of all study image data collection for all participants [approximately 1 year]
  The sensitivity of FFNP PET /MR is defined as the ability of readers (radiologists) to correctly detect areas that will respond to treatment, as determined by histopathologic evaluation.
Specificity of 18F-fluorofuranylnorprogesterone (FFNP) PET/MRI for predicting response to progestin therapy in CAH /EC patients | Upon completion of all study image data collection for all participants [approximately 1 year]
  The specificity is similarly defined as the ability of readers to determine areas that will fail to respond to treatment, as determined by histopathologic evaluation.

SECONDARY OUTCOMES:
Correlate FFNP Mean Standardized Uptake Value (SUVmean) at baseline and on repeat examination with estrogen and progesterone receptor expression in the CAH/EC tissues at baseline and after 6 months of treatment. | Upon completion of all study image data collection for all participants [approximately 1 year]
  The association between SUVmean and tumor volume and the degree of estrogen/progesterone receptor will be evaluated using random coefficient trajectory models, separately for each outcome. These models allow a separate outcome trajectory for each patient, accounting for within-patient correlations arising from the fact that measurements are taken at multiple timepoints. Estrogen/progesterone receptor will be included as a fixed effect, along with the interaction of this fixed effect and time. A p-value <0.05 for this interaction will be considered evidence that the association between the outcome and estrogen/progesterone receptor varies by time. A patient-level random intercept will be included in the models. Differences in predicted means of the outcomes at each time point will be computed and tested to see if they differ from 0; p-values <0.05 for these tests will be considered evidence of a difference in predicted means by estrogen/progesterone values.
Correlate FFNP Maximum Standardized Uptake Value (SUVmax) at baseline and on repeat examination with estrogen and progesterone receptor expression in the CAH/EC tissues at baseline and after 6 months of treatment. | Upon completion of all study image data collection for all participants [approximately 1 year]
  The association between SUVmax and tumor volume and the degree of estrogen/progesterone receptor will be evaluated using random coefficient trajectory models, separately for each outcome. These models allow a separate outcome trajectory for each patient, accounting for within-patient correlations arising from the fact that measurements are taken at multiple timepoints. Estrogen/progesterone receptor will be included as a fixed effect, along with the interaction of this fixed effect and time. A p-value <0.05 for this interaction will be considered evidence that the association between the outcome and estrogen/progesterone receptor varies by time. A patient-level random intercept will be included in the models. Differences in predicted means of the outcomes at each time point will be computed and tested to see if they differ from 0; p-values <0.05 for these tests will be considered evidence of a difference in predicted means by estrogen/progesterone values.

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Oldan, MD, Principal Investigator — University of North Carolina, Chapel Hill

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with the University of North Carolina (UNC).
Supporting Information: Study Protocol
Time Frame: 9 to 36 months following publication
Access Criteria: The investigator who proposes to use the data has approval from an IRB, IEC, or REB, as applicable, and an executed data use/sharing agreement with UNC.